CLINICAL TRIAL: NCT02623322
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Trial of MHAA4549A, a Monoclonal Antibody, Administered as Monotherapy for the Treatment of Acute Uncomplicated Seasonal Influenza A Infection in Otherwise Healthy Adults
Brief Title: A Study of MHAA4549A as Monotherapy for Acute Uncomplicated Seasonal Influenza A in Otherwise Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GV29893; 2016-000425-40 (EudraCT Number)
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Influenza A
MeSH Terms: interventions — gedivumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MHAA4549A 3600 milligrams (mg) (Experimental): Participants will receive single-dose MHAA4549A, 3600 mg, by intravenous (IV) administration.
  Interventions: Drug: MHAA4549A
- MHAA4549A 8400 mg (Experimental): Participants will receive single-dose MHAA4549A, 8400 mg, by IV administration.
  Interventions: Drug: MHAA4549A
- Placebo (Placebo Comparator): Participants will receive single-dose placebo by IV administration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MHAA4549A — MHAA4549A will be administered as a single dose by IV administration.
  Arms: MHAA4549A 3600 milligrams (mg); MHAA4549A 8400 mg
Drug: Placebo — Placebo will be administered as a single dose by IV administration.
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled single dose study in otherwise healthy adults with acute uncomplicated seasonal influenza A to assess the safety and tolerability, efficacy, and pharmacokinetics of MHAA4549A.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy participants
* Positive test for influenza A infection
* No more than 72 hours elapsed between onset of influenza-like illness and start of study drug
* Presence of at least one moderate or severe constitutional symptom such as headache, myalgia, fever, chills, fatigue, anorexia, or nausea PLUS one moderate or severe respiratory symptom such as cough, sore throat, or rhinorrhea
* For women of childbearing potential: negative pregnancy test and agreement to use acceptable contraceptive methods for at least 120 days after study drug administration
* For men: agreement to use acceptable contraceptive methods for at least 30 days after study drug administration

Exclusion Criteria:

* Creatinine clearance less than or equal to (</=) 80 milliliters per minute (mL/min)
* Any significant medical conditions or laboratory abnormalities
* Clinical signs and symptoms consistent with otitis, bronchitis, sinusitis, or pneumonia or active bacterial infection
* Use of antiviral therapy in the period from onset of influenza-like illness and prior to enrollment
* Pregnancy at Screening or is currently pregnant or breastfeeding
* Investigational therapy within 30 days or 5 half-lives prior to start of study drug, whichever is greater
* Prior anti-influenza monoclonal antibody use
* Receipt of a nasal influenza A vaccine within 14 days prior to Screening
* Positive test for influenza B or influenza A+B within 2 weeks prior to study drug
* History of significant tobacco use or drug/alcohol abuse
* Chronic use of oral or inhaled corticosteroids within 30 days prior to Screening
* Autoimmune disease, known immunodeficiency of any cause, or use of immunosuppressive medications
* History of any chronic respiratory condition
* Human immunodeficiency virus (HIV) with cluster of differentiation (CD) 4 count </= 200 cells per milliliter (cells/mL) in the past 12 months
* Serious infection requiring oral or IV antibiotics within 14 days prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (80):
- United States (38):
  - North Alabama Research Center LLC, Athens, Alabama
  - WCCT Global, LLC, Costa Mesa, California
  - Lalla-Reddy Medical Corporation, Fountain Valley, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Integrity Clinical Research, Doral, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - The Community Research Of South Florida, Hialeah, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Oceane7 Clinical Research, Miami, Florida
  - Central Florida Internists, Saint Cloud, Florida
  - Tampa General Hospital, Tampa, Florida
  - Advanced Research Institute, Inc., Trinity, Florida
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Professional Research Network of Kansas, Wichita, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Kentucky Lung Clinic, Hazard, Kentucky
  - MedPharmics, Metairie, Louisiana
  - Acadiana Medicine Clinic, Opelousas, Louisiana
  - Anne Arundel Medical Center; Anne Arundel Health System, Annapolis, Maryland
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - Sinai Grace Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Barnes Jewish Hospital, St Louis, Missouri
  - Mercury Street Medical Group, Butte, Montana
  - Barrett Clinic, P.C., La Vista, Nebraska
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - Wake Research Associates, Raleigh, North Carolina
  - Center For Medical Research LLC, Providence, Rhode Island
  - Emergency MD, Boiling Springs, South Carolina
  - HCCA Clinical Research Solutions, Franklin, Tennessee
  - Clinical Research Solutions PC, Knoxville, Tennessee
  - Clinical Research Solutions, LLC, Smyrna, Tennessee
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Centex Studies, Houston, Texas
  - Centex Studies, Pharr, Texas
- Canada (5):
  - Manna Research Vancouver, Vancouver, British Columbia
  - Moncton Hospital, Moncton, New Brunswick
  - Manna Research, Toronto, Ontario
  - Q and T Research, Gatineau, Quebec
  - inVentiv Health Clinique, Québec
- New Zealand (4):
  - Henderson Medical Centre, Auckland
  - Optimal Clinical Trials, Auckland
  - RMC Medical Research Ltd, Dunedin
  - Tauranga Hospital, Tauranga
- South Africa (17):
  - Johese Clinical Research, Centurion
  - Durban International Clinical Research Site, Durban
  - Vawda Z Private Practice, Durban
  - Dr Peter John Sebastian; Dr PJ Sebastian, Durban
  - Into Research; Life Groenkloof Hospital Medical Centre, Groenkloof
  - Worthwhile Clinical Trials, Johannesburg
  - Newtown Clinical Research, Johannesburg
  - Clinresco Centres (Pty) Ltd, Kempton Park
  - Peermed Clinical Trial Centre, Kempton Park
  - Klerksdorp /Tshepong Hospital Complex, Klerksdorp
  - DJW Navorsing, Krugersdorp
  - I Engelbrecht Research, Lyttleton
  - Syzygy Clinical Research; Unit 3 to 7, Pretoria Gauteng Province
  - Jongaie Research, Pretoria West
  - Queenswood CTC, Queenswood
  - Wits Clinical Research, Soweto
  - Welkom Clinical Trial Centre, Welkom
- South Korea (7):
  - Hallym University Sacred Heart Hospital, Anyang-si
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Gachon University Gil Hospital, Incheon
  - Korea University Anam Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Wonju Christian Hospital, Wŏnju
- Spain (6):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Mutua de Terrassa; Servicio de Oncologia, Terrassa, Barcelona
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital de Galdakao, Galdacao, Vizcaya
  - Hospital del Mar, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
- United Kingdom (3):
  - Surrey Clinical Research Centre; University of Surrey, Guildford
  - Barts and the London NHS Trust., London
  - The James Cook University Hospital, Middlesbrough

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 34 investigational sites in 6 countries including the United States (15 centers), South Africa (12 centers), Canada, Spain, New Zealand (2 centers in each country), and Great Britain (1 center).
Pre-assignment Details: Randomization was stratified by onset of influenza-like illness (≤ 36 hours and > 36 hours) and a permuted block randomization method was used to obtain an approximate 1:1:1 ratio of subjects in the 3600 mg MHAA4549A, 8400 mg MHAA4549A, and placebo strata.
Groups:
- Placebo: Participants received single-dose placebo by intravenous (IV) administration.
- MHAA4549A 3600 mg: Participants received single-dose MHAA4549A, 3600 milligrams (mg), by IV administration.
- MHAA4549A 8400 mg: Participants received single-dose MHAA4549A, 8400 mg, by IV administration.
Period: Overall Study
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Started | 43 | 41 | 40
Completed | 41 | 40 | 40
Not Completed | 2 | 1 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population included all participants randomized to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg | Total
Number analyzed (Participants) | 43 | 41 | 40 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (10.8) | 36.5 (12.5) | 35.0 (13.6) | 37.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 22 | 71
  Male | 16 | 19 | 18 | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 7
  Not Hispanic or Latino | 40 | 38 | 38 | 116
  Not Stated | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 4 | 1 | 7
  Black or African American | 13 | 7 | 15 | 35
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 0 | 3
  White | 27 | 26 | 23 | 76
  Multiple | 0 | 0 | 1 | 1
  Unknown | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not considered related to the study drug.
Time Frame: Baseline to Day 100
Population: The safety population included all participants randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 43 | 41 | 40
percentage of participants | 30.2 | 39.0 | 30.0

2. Secondary Outcome: Percentage of Participants Requiring Hospitalization for Influenza-Related Complications
Time Frame: Baseline to Day 100
Population: The intent-to-treat infected (ITTI) population included all randomized participants who had an influenza A infection confirmed by central polymerase chain reaction (PCR).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 33 | 35 | 31
percentage of participants | 0 | 0 | 0

3. Secondary Outcome: Duration of Hospitalization for Influenza-Related Complications
Time Frame: Baseline to Day 100
Population: as for outcome 2
Measure: Number; unit: days
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 33 | 35 | 31
days | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants Requiring Antibiotics for Secondary Bacterial Respiratory Infections
Description: Participants with antibiotic usage for secondary bacterial respiratory infections were identified by counting participants with AEs containing the terms, "pneumonia, lung, myocarditis, ARDS (acute respiratory distress syndrome), otitis media, or respiratory."
Time Frame: Baseline to Day 100
Population: The intent-to-treat infected (ITTI) population included all randomized participants who had an influenza A infection confirmed by central PCR.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 33 | 35 | 31
percentage of participants | 3.0 [0.32 to 11.28] | 0 [0.00 to 6.37] | 0 [0.00 to 7.16]
Statistical Analysis 1: Comparison: Placebo vs MHAA4549A 3600 mg; Test type: Superiority; p = 0.3031, Cochran-Mantel-Haenszel; Difference in event rates (Wald) = -3.03, 80% CI 2-sided [-12.25 to 6.19]
Statistical Analysis 2: Comparison: Placebo vs MHAA4549A 8400 mg; Test type: Superiority; p = 0.3324, Cochran-Mantel-Haenszel; Difference in event rates (Wald) = -3.03, 80% CI 2-sided [-12.82 to 6.76]

5. Secondary Outcome: Percentage of Participants With Complications of Influenza
Description: Participants with complications of influenza were identified by counting participants with AEs containing the terms, "pneumonia, lung, myocarditis, ARDS (acute respiratory distress syndrome), otitis media, or respiratory."
Time Frame: Baseline to Day 100
Population: ITTI population included all randomized participants who had an influenza A infection confirmed by central PCR.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 33 | 35 | 31
percentage of participants | 3.0 [0.32 to 11.28] | 0 [0.00 to 6.37] | 0 [0.00 to 7.16]
Statistical Analysis 1: Comparison: Placebo vs MHAA4549A 3600 mg; Test type: Superiority; p = 0.3031, Cochran-Mantel-Haenszel; Difference in event rates (Wald) = -3.03, 80% CI 2-sided [-12.25 to 6.19]
Statistical Analysis 2: Comparison: Placebo vs MHAA4549A 8400 mg; Test type: Superiority; p = 0.3324, Cochran-Mantel-Haenszel; Difference in event rates (Wald) = -3.03, 80% CI 2-sided [-12.82 to 6.76]

6. Secondary Outcome: Percentage of Participants With Influenza A Relapse/Reinfection
Time Frame: Baseline to Day 100
Population: ITTI population included all randomized participants who had an influenza A infection confirmed by central PCR.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 33 | 35 | 31
percentage of participants | 0 | 0 | 0

7. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) of MHAA4549A
Description: The AUC is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption. AUC was measured in micrograms times hours per milliliter (mcg*h/mL).
Time Frame: Up to Day 100 (collections scheduled pre-dose [0 hours]; 60 minutes post-dose; and on Days 3, 5, 7, 30, and 100 post-dose; infusion duration = 2 hours)
Population: Data were collected for this outcome measure.
Arm/Group | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of MHAA4549A
Time Frame: as for outcome 7
Population: The pharmacokinetic (PK)-evaluable population included all participants who received MHA4549A.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 40 | 37
mcg/mL | 1050 (299) | 2190 (581)

9. Secondary Outcome: Time to Alleviation of Symptoms of Influenza A Infection
Description: Time to alleviation of all 7 symptoms (i.e., nasal congestion, sore throat, cough, aches, fatigue, headaches, chills/sweats) was assessed using a rating scale of 0 (none), 1 (mild), 2 (moderate), or 3 (severe) for each symptom. The outcome was defined in two ways: time to a total symptom score of <=1 and time to a total symptom score of <=7. Resolution had to be maintained for 24 hours without use of symptom relief medications. For participants who were enrolled with mild symptoms, the symptom score had to be reduced by one point during the study duration.
Time Frame: Baseline to Day 14
Population: ITTI population included all randomized participants who had an influenza A infection confirmed by central PCR. Data are reported for evaluable participants.
Measure: Median (80% Confidence Interval); unit: hours
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 33 | 35 | 31
hours
  Total Symptom Score of <=1 | 117.30 [108.62 to 157.15] | 153.80 [125.52 to 175.23] | 145.82 [132.98 to 156.68]
  Total Symptom Score of <=7: number analyzed (Participants) | 33 | 34 | 31
  Total Symptom Score of <=7 | 44.50 [27.23 to 58.65] | 74.18 [64.32 to 87.98] | 65.59 [44.12 to 87.23]
Statistical Analysis 1: Comparison: Placebo vs MHAA4549A 3600 mg; Total Symptom Score of <=1; Test type: Superiority; p = 0.7858, Wilcoxon; Hazard Ratio (HR) = 0.92, 80% CI 2-sided [0.62 to 1.37]
Statistical Analysis 2: Comparison: Placebo vs MHAA4549A 8400 mg; Total Symptom Score of <=1; Test type: Superiority; p = 0.5170, Wilcoxon; Hazard Ratio (HR) = 0.90, 80% CI 2-sided [0.59 to 1.36]
Statistical Analysis 3: Comparison: Placebo vs MHAA4549A 3600 mg; Total Symptom Score of <=7; Test type: Superiority; p = 0.0312, Wilcoxon; Hazard Ratio (HR) = 0.63, 80% CI 2-sided [0.45 to 0.89]
Statistical Analysis 4: Comparison: Placebo vs MHAA4549A 8400 mg; Total Symptom Score of <=7; Test type: Superiority; p = 0.2044, Wilcoxon; Hazard Ratio (HR) = 0.74, 80% CI 2-sided [0.53 to 1.04]

10. Secondary Outcome: Percentage of Participants With Influenza-Related Deaths
Time Frame: Baseline to Day 100
Population: The safety population included all participants randomized to treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
Number analyzed (Participants) | 43 | 41 | 40
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Day 100
Description: The safety population included all participants randomized to treatment.
Arm/Group | Placebo | MHAA4549A 3600 mg | MHAA4549A 8400 mg
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/41 | 1/40
Other Adverse Events (participants affected / at risk) | 4/43 | 7/41 | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | MHAA4549A 3600 mg (N=41) | MHAA4549A 8400 mg (N=40)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | MHAA4549A 3600 mg (N=41) | MHAA4549A 8400 mg (N=40)
Nausea (Gastrointestinal disorders) | 2 | 3 | 3
Bronchitis (Infections and infestations) | 1 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/22/NCT02623322/Prot_SAP_000.pdf